CLINICAL TRIAL: NCT05517226
Title: A Phase I, Parallel-group, Multi-center, Open-label, Investigation of the Pharmacokinetics, Safety and Tolerability of a Single Subcutaneous Injection of Cotadutide in Participants With Mild, Moderate or Severe Hepatic Impairment Compared to Participants With Normal Hepatic Function
Brief Title: Pharmacokinetics of Cotadutide in Participants With Hepatic Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Discontinuing the development of cotadutide, a daily injectable GLP-1/glucagon co-agonist, is based on strategic pipeline considerations.
  The premature closure is not due to any newly observed safety signals or a change in the risk/benefit profile.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5671C00008
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Hepatic Impairment
Keywords: Cotadutide; Hepatic impairment
MeSH Terms: interventions — cotadutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Participants in each cohort will receive Dose A cotadutide subcutaneously.
  Interventions: Combination Product: Cotadutide
- Cohort 2 (Experimental): Participants in each cohort will receive Dose A cotadutide subcutaneously.
  Interventions: Combination Product: Cotadutide
- Cohort 3 (Experimental): Participants in each cohort will receive Dose A cotadutide subcutaneously.
  Interventions: Combination Product: Cotadutide
- Cohort 4 (Experimental): Participants in each cohort will receive Dose A cotadutide subcutaneously.
  Interventions: Combination Product: Cotadutide

INTERVENTIONS:
Combination Product: Cotadutide — Participants will receive cotadutide subcutaneously.

SUMMARY:
This study will assess the pharmacokinetics (PK), safety, and tolerability of a single subcutaneous injection of cotadutide in participants with mild, moderate or severe hepatic impairment compared to participants with normal hepatic function.

DETAILED DESCRIPTION:
This study will consist of four cohorts (Cohort 1, Cohort 2, Cohort 3, and Cohort 4).

Participants will be assigned to each of the cohorts as per Child-Pugh classification:

* Cohort 1: Mild hepatic impairment (Child-Pugh A), cotadutide 50 μg
* Cohort 2: Moderate hepatic impairment (Child-Pugh B), cotadutide 50 μg
* Cohort 3: Severe hepatic impairment (Child-Pugh C), cotadutide 50 μg
* Cohort 4: Normal hepatic function, cotadutide 50 μg

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 to ≤ 85 years of age at the time of signing the Informed Consent Form (ICF).
* Body mass index ≥ 18 kg/m2 to < 40 kg/m2.
* Female participants of childbearing potential must use at least one highly effective form of birth control.
* Capable of giving signed informed consent.

Participants with hepatic impairment only

- Diagnosis of chronic (≥ 6 months) and stable hepatic impairment (eg, no clinically significant change in signs, symptoms, or laboratory parameters of hepatic disease status within 30 days prior to study Screening).

Exclusion Criteria:

All participants

* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to cotadutide.
* Any clinically important abnormalities in rhythm, conduction or morphology of the 12-lead resting electrocardiogram (ECG) and any clinically important abnormalities in the 12-lead ECG as considered by the Investigator that may interfere with the interpretation of QT interval corrected for heart rate using Fridericia's formula (QTcF), including abnormal ST-T-wave morphology, or left ventricular hypertrophy

  1. Prolonged QTcF > 470 ms or family history of long QT syndrome.
  2. PR (PQ) interval shortening < 120 ms.
  3. PR (PQ) interval prolongation (> 220 ms) intermittent or permanent second or third degree atrioventricular (AV) block, or AV dissociation.
  4. Persistent or intermittent complete bundle branch block, or intraventricular conduction delay with QRS > 119 ms.
* Any evidence of additional severe or uncontrolled systemic disease or laboratory finding that makes it unsafe for the participant to participate in the study.
* Impaired renal function, defined as estimated glomerular filtration rate (eGFR) < 30 mL/minute/1.73 m2 at Screening.
* Any positive result on Screening for serum hepatitis B surface antigen, anti-Core HBV antibody, hepatitis C antibody, or human immunodeficiency virus (HIV).
* Any sign and confirmation of coronavirus disease 2019 (COVID19) infection:
* Participants with concurrent or previous use of a glucagon-like peptide-1 (GLP1) receptor agonist.
* Use of prohibited prescribed or nonprescribed medication during the 2 weeks prior to the first administration of Investigational Medicinal Product (IMP) or longer if the medication has a long half-life.
* History of neoplastic disease within 5 years prior to Screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer.
* Presence of hepatocellular carcinoma or acute liver disease caused by an infection or drug toxicity.

Participants with hepatic impairment only

* Severe portal hypertension or surgical porto-systemic shunts.
* Biliary obstruction or other causes of hepatic impairment not related to parenchymal disorder and/or disease of the liver.
* Clinically relevant hepatic encephalopathy.
* Severe ascites defined as ascites requiring paracentesis and albumin at 4-week intervals or less.
* Fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within the 28-day Screening period.
* Post liver transplantation.
* Platelet count < 50 × 109/L and/or neutrophil count < 1.2 × 109/L and/or hemoglobin < 8.5 g/dL or INR >2.3.

Participants with normal hepatic function only

* History or presence of hepatic disease or evidence of other known forms of known chronic liver disease.
* History or presence of gastrointestinal, hepatic, or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Urinary albumin-to-creatinine ratio > 3 mg/μmol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma (peak) drug concentration [Cmax] | Day 1 to Day 3
  The Cmax of a single dose of cotadutide in participants with mild, moderate, or severe hepatic impairment compared to those with normal hepatic function will be assessed.
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 to Day 3
  The AUCinf of a single dose of cotadutide in participants with mild, moderate, or severe hepatic impairment compared to those with normal hepatic function will be assessed.
Area under the plasma concentration-curve from time zero to last quantifiable concentration (AUClast) | Day 1 to Day 3
  The AUClast of a single dose of cotadutide in participants with mild, moderate, or severe hepatic impairment compared to those with normal hepatic function will be assessed.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Day 1 to Day 3
  The tmax of a single dose of cotadutide in participants with mild, moderate, or severe hepatic impairment compared to those with normal hepatic function will be assessed.
Terminal half-life (t½λz) | Day 1 to Day 3
  The t½λz of a single dose of cotadutide in participants with mild, moderate, or severe hepatic impairment compared to those with normal hepatic function will be assessed.
Apparent total body clearance (CL/F) | Day 1 to Day 3
  The CL/F of a single dose of cotadutide in participants with mild, moderate, or severe hepatic impairment compared to those with normal hepatic function will be assessed.
Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1 to Day 3
  The Vz/F of a single dose of cotadutide in participants with mild, moderate, or severe hepatic impairment compared to those with normal hepatic function will be assessed.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From time of first dose to the final follow-up visit (Day 29)
  The safety, and tolerability of a single dose of cotadutide in participants with hepatic impairment will be assessed.
Incidence of ADAs (anti-drug antibodies) | From time of first dose to the final follow-up visit (Day 29)
  The safety, and tolerability of a single dose of cotadutide in participants with hepatic impairment will be assessed.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Hialeah, Florida
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home